CLINICAL TRIAL: NCT05891262
Title: A Phase 1, Single-center, Open-label, Single-sequence Study to Evaluate the Drug-drug Interaction Potential of BMS-986196 With Oral Contraceptives in Healthy Female Participants
Brief Title: A Study to Evaluate the Drug-drug Interaction of BMS-986196 With Oral Contraceptives in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM038-023
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Healthy Female Volunteers
Keywords: Pharmacokinetics; BMS-986196; Hormonal contraceptives; Ethinyl estradiol; Norethindrone; Female volunteers
MeSH Terms: interventions — norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination; Ethinyl Estradiol; Norethindrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BMS-986196 and Loestrin (Experimental)
  Interventions: Drug: BMS-986196; Drug: Loestrin

INTERVENTIONS:
Drug: BMS-986196 — Specified dose on specified days
Drug: Loestrin — Specified dose on specified days
  Other Names: Ethinyl estradiol (EE) and norethindrone (NET)

SUMMARY:
The purpose of this study is to evaluate the effect of BMS-986196 when coadministered with combined hormonal oral contraceptives (ethinyl estradiol [EE] and norethindrone [NET]) in healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be genetically and hormonally female with intact ovarian function by medical history/menstrual cycles.
* Body mass index between 18.0 and 35.0 kilograms/meter square (kg/m^2), inclusive, at screening.
* Healthy female participants as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluations.

Exclusion Criteria:

* Any significant acute or chronic medical illness judged to be clinically significant by the investigator and/or Sponsor Medical Monitor.
* History of clinically significant heart disease, including ischemia, infarction, clinically significant arrhythmias, sinus syndrome, hypertension, clinically significant ECG abnormalities, venous thromboembolism, or any congenital heart disease (as assessed by the investigator).
* Current or recent (within 3 months of study intervention administration) gastrointestinal disease that could possibly affect drug absorption, distribution, metabolism and excretion (for example, bariatric procedure).
* Any major surgery within 4 weeks of study intervention administration, including gastrointestinal surgery that could affect the absorption of study intervention.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | At Day 1 and Day 20
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | At Day 1 and Day 20
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC [INF]) | At Day 1 and Day 20

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | At Day 1 and Day 20
Terminal half-life (T-HALF) | At Day 1 and Day 20
Apparent total body clearance (CLT/F) | At Day 1 and Day 20
Number of participants with Adverse Events (AEs) | Up to Day 49
Number of participants with Serious AEs (SAEs) | Up to Day 49
Number of participants with clinical laboratory abnormalities | Up to Day 49
Number of participants with vital sign abnormalities | Up to Day 49
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 49
Number of participants with physical examination abnormalities | Up to Day 49
Number of participants with any abnormal columbia-suicide severity rating scale (C-SSRS) | Up to Day 49

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Altasciences, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com